CLINICAL TRIAL: NCT05457634
Title: Nicotine Uptake and Abuse Liability Assessments of 5 Blu Disposable Electronic Cigarettes in Comparison to a Combustible Cigarette
Brief Title: Nicotine Uptake and Abuse Liability Assessments of Blu Disposable Electronic Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fontem US LLC (Industry)
Responsible Party: Sponsor
Organization: Fontem Ventures BV (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Fontem-PK-01
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- blu Disposable Flavor A (Experimental): Subjects who use the blu disposable electronic cigarette 2.4% nicotine with Flavor A
  Interventions: Other: blu Disposable A
- blu Disposable Flavor B (Experimental): Subjects who use the blu disposable electronic cigarette 2.4% nicotine with Flavor B
  Interventions: Other: blu Disposable B
- blu Disposable Flavor C (Experimental): Subjects who use the blu disposable electronic cigarette 2.4% nicotine with Flavor C
  Interventions: Other: blu Disposable C
- blu Disposable Flavor D (Experimental): Subjects who use the blu disposable electronic cigarette 2.4% nicotine with Flavor D
  Interventions: Other: blu Disposable D
- blu Disposable Flavor E (Experimental): Subjects who use the blu disposable electronic cigarette 2.4% nicotine with Flavor E
  Interventions: Other: blu Disposable E
- Combustible cigarette (Active Comparator): Subjects who use their own brand of combustible cigarette
  Interventions: Other: Combustible Cigarette

INTERVENTIONS:
Other: Combustible Cigarette — Subjects smoke their Usual Brand Combustible Cigarette, for 2 consecutive product use sessions. 1. Defined session: 10 puffs, each 30 seconds apart. 2. Ad libitum session: 60 minutes ad-libitum use.
  Arms: Combustible cigarette
Other: blu Disposable A — Subjects use the blu disposable e-cigarette with flavor A, 2.4% nicotine, for 2 consecutive product use sessions. 1. Defined session: 10 puffs, each 30 seconds apart. 2. Ad libitum session: 60 minutes ad-libitum use.
  Arms: blu Disposable Flavor A
Other: blu Disposable B — Subjects use the blu disposable e-cigarette with flavor B, 2.4% nicotine, for 2 consecutive product use sessions. 1. Defined session: 10 puffs, each 30 seconds apart. 2. Ad libitum session: 60 minutes ad-libitum use.
  Arms: blu Disposable Flavor B
Other: blu Disposable C — Subjects use the blu disposable e-cigarette with flavor C, 2.4% nicotine, for 2 consecutive product use sessions. 1. Defined session: 10 puffs, each 30 seconds apart. 2. Ad libitum session: 60 minutes ad-libitum use.
  Arms: blu Disposable Flavor C
Other: blu Disposable D — Subjects use the blu disposable e-cigarette with flavor D, 2.4% nicotine, for 2 consecutive product use sessions. 1. Defined session: 10 puffs, each 30 seconds apart. 2. Ad libitum session: 60 minutes ad-libitum use.
  Arms: blu Disposable Flavor D
Other: blu Disposable E — Subjects use the blu disposable e-cigarette with flavor E, 2.4% nicotine, for 2 consecutive product use sessions. 1. Defined session: 10 puffs, each 30 seconds apart. 2. Ad libitum session: 60 minutes ad-libitum use.
  Arms: blu Disposable Flavor E

SUMMARY:
This study assesses the nicotine uptake, abuse liability and puffing topography of blu disposable e-cigarettes in adult combustible cigarette smokers. Nicotine uptake, subjective effects, and puff topography are evaluated and compared with subjects' usual brand combustible cigarette.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be current smokers (≥10 per day) of combustible cigarettes for at least 6 continuous months before Visit 1 and may be occasional users of e-cigarettes
* Subjects have urine cotinine >200 ng/mL and exhaled carbon monoxide > 10 ppm at Screening
* Subject has a seated systolic blood pressure ≤160 mmHg, diastolic blood pressure

  ≤95 mmHg, and heart rate ≤100 bpm
* Females of childbearing potential who are practicing a reliable method of contraception

Exclusion Criteria:

* Subjects who have used any nicotine or tobacco product other than e-cigarettes or combustible cigarettes in the 14 days prior to Visit 1
* Subjects who have an acute illness requiring treatment in the 4 weeks prior to Visit 1
* Subjects with clinically significant and relevant abnormalities of medical history.
* Subjects who have used any prescription or over-the-counter smoking cessation treatments within 30 days prior to Visit 1
* Pregnant or breastfeeding female subjects

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Nicotine Cmax0-120 | 5 minutes before and at 3, 5, 7, 10, 15, 20, 30, 45, 60, 90, and 120 minutes after the first puff
  Maximum plasma nicotine concentration, during the defined use session, adjusted for baseline nicotine
Nicotine Cmax120-180 | at 15, 30, 45, and 60 minutes after the start of the ad libitum use session (ad libitum session starts at 120 min relative to first puff of controlled use session)
  Maximum plasma nicotine concentration during the ad libitum use session, adjusted for baseline nicotine
Nicotine AUC0-120 | 5 minutes before and at 3, 5, 7, 10, 15, 20, 30, 45, 60, 90, and 120 minutes after the first puff
  Area under the plasma nicotine concentration-time curve from time 0 to 120 minutes during the defined use session
Nicotine AUC120-180 | at 15, 30, 45, and 60 minutes after the start of the ad libitum use session
  Area under the plasma nicotine concentration-time curve from time 120 minutes to 180 minutes, i.e. during the ad libitum use session
Urge to Smoke - Defined use | 5 minutes before and at 3, 5, 7, 10, 15, 20, 30, 45, 60, 90, and 120 minutes after the first puff
  Subjects answer "How strong is your current urge to smoke your usual brand cigarette?" on a Visual Analog Scale: from "No Urge" at the left to "Very Strong Urge" at the right.
Urge to Smoke - Ad libitum use | at 15, 30, 45, and 60 minutes after the start of the ad libitum use session
  Subjects answer "How strong is your current urge to smoke your usual brand cigarette?" on a Visual Analog Scale: from "No Urge" at the left to "Very Strong Urge" at the right.

SECONDARY OUTCOMES:
Puff topography: puff count | Throughout ad libitum use session (60 minutes)
  Measured during the ad libitum use session with a CReSS Pocket topography device

OTHER OUTCOMES:
Safety Outcome: heart rate after defined use | At 8 minutes relative to first puff of defined use session
  Heart rate after the subject has spent at least 5 minutes in the seated position
Safety Outcome: heart rate after ad libitum use | At 60 minutes relative to first puff of ad libitum use session
  Heart rate after the subject has spent at least 5 minutes in the seated position
Safety Outome: systolic blood pressure after defined use | At 8 minutes relative to first puff of defined use session
  Blood pressure measured after the subject has spent at least 5 minutes in the seated position
Safety Outome: systolic blood pressure after ad libitum use | At 60 minutes relative to first puff of ad libitum use session
  Blood pressure measured after the subject has spent at least 5 minutes in the seated position
Safety Outome: diastolic blood pressure after defined use | At 8 minutes relative to first puff of defined use session
  Blood pressure measured after the subject has spent at least 5 minutes in the seated position
Safety Outome: diastolic blood pressure after ad libitum use | At 60 minutes relative to first puff of ad libitum use session
  Blood pressure measured after the subject has spent at least 5 minutes in the seated position

CONTACTS AND LOCATIONS:
Locations (1):
- LA Clinical Trials, LLC, Burbank, California, United States

DOCUMENTS (2):
  • Study Protocol (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT05457634/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT05457634/SAP_001.pdf